CLINICAL TRIAL: NCT00426894
Title: Longitudinal Microbial Surveillance in Children Hospitalized for Cardiac Surgery Before the Operation and During Hospitalization
Brief Title: Microbial Surveillance in Children Hospitalized for Cardiovascular Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: yael01-HMO-CTIL
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2007-01

CONDITIONS: Cardiac Surgery; Perioperative Prophylaxis
Keywords: surveillance cultures; children; cardiac surgery; perioperative prophylaxis

INTERVENTIONS:
Procedure: samples from nostrils, mouth, axillas, perianal area and postoperative wound

SUMMARY:
the purpose of this study is to determine whether children who are hospitalised waiting for cardiac surgery for several days in pediatric or pediatric surgery department acquire resistant microbial flora, thus necessitating broad spectrum antibiotics for perioperative prophylaxis.

DETAILED DESCRIPTION:
Background

Guidelines for antimicrobial prophylaxis for cardiac surgery advise using first generation cephalosporin for those children coming from home. Large number of children that pass cardiac surgery in Hadassah University Hospital, Jerusalem, are hospitalized for several days before the operation in Pediatric Surgery department due to administrative reasons. These children receive broad spectrum antibiotics, vancomycin and ceftazidime, as a peri-operative prophylaxis, in order to prevent infection with hospital acquired flora with which they could become colonized with during this period. This policy causes exposure to broad spectrum antibiotics from the beginning in these children, and also providing an antimicrobial pressure in the intensive care unit, influencing the development of resistant flora.

There is no documentation that these children acquire resistant flora during there hospitalization in the pre-operative period. We suggest checking microbial flora in those children hospitalized for cardiac surgery, in order to determine the need for broad spectrum antimicrobial prophylaxis.

Goals

To check microbial flora in children hospitalized for cardiac surgery on different time points: on admission and during hospitalization in Pediatric Surgery Department, on admission to PICU (immediately after operation),after 3 - 5 days,when drains are extracted.

To document if there is a change in resistance pattern of microbial pathogens during these periods

To determine the optimal regimen for antimicrobial prophylaxis for those children who need to be hospitalized in this department before the operation

Methods

Surveillance cultures would be taken from children who are hospitalized for cardiac surgery on several time points:

1. on admission to Pediatric Surgery or other department pre-operatively
2. once weekly afterwards, if they continue to be hospitalized without surgery
3. on admission to PICU after surgery
4. during their subsequent hospitalization in PICU after 3 - 5 days
5. on the day of drains extraction

These cultures will include the cultures of nostrils, throat,axillas, perineum and rectum and post operative wound.

ELIGIBILITY:
Inclusion Criteria:

* All children and infants who are hospitalized in general pediatrics or pediatric surgery department before they undergo cardiac surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Dina Averbuch, MD, Principal Investigator — Hadassah University Hospital, Jerusalem, Israel
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Background] Bratzler DW, Houck PM; Surgical Infection Prevention Guideline Writers Workgroup. Antimicrobial prophylaxis for surgery: an advisory statement from the National Surgical Infection Prevention Project. Am J Surg. 2005 Apr;189(4):395-404. doi: 10.1016/j.amjsurg.2005.01.015. PMID 15820449